CLINICAL TRIAL: NCT04214782
Title: Detection of Ovarian Cancer Using an Artificial Intelligence Enabled Transvaginal Ultrasound Imaging Algorithm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Hubei Cancer Hospital (Other); Qilu Hospital of Shandong University (Other); Henan Cancer Hospital (Other Government); Xiangyang Central Hospital (Other); The First People's Hospital of Jingzhou (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2019-TJ-OVAB
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transvaginal Ultrasound diagnosis (No Intervention): radiologists interpretTransvaginal Ultrasound images without the help of Artificial Intelligence (AI) algorithm
- AI enabled Transvaginal Ultrasound diagnosis (Experimental): radiologists interpretTransvaginal Ultrasound images with the help of Artificial Intelligence algorithm
  Interventions: Diagnostic Test: Artificial Intelligence Enabled Transvaginal Ultrasound Imaging algorithm

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence Enabled Transvaginal Ultrasound Imaging algorithm — AI Enabled Transvaginal Ultrasound diagnosis for ovarian cancer
  Other Names: AI Enabled Transvaginal Ultrasound diagnosis
  Arms: AI enabled Transvaginal Ultrasound diagnosis

SUMMARY:
Ovarian cancer is relatively rare but fatal with an annual incidence rate of 11.8 per 100 000 and a high mortality-to-incidence ratio of >0.6. The modest diagnostic accuracy of TVU has risen some concerns about the over-treatment.Now, with the development of artificial intelligence (AI), we may have a better chance to interpret TVU imagines with high efficiency, reproducibility and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for Transvaginal Ultrasound examination for adnexal lesions;
* Women aged over 18 years old;
* Women willing to participant in this study evidenced by signing the informed consent.

Exclusion Criteria:

* Women without adnexa for any reasons at the time of Transvaginal Ultrasound examination, including but not limited to receiving surgical removal for adnexa;
* Women with a pathologic diagnosis of ovarian cancer before the Transvaginal Ultrasound examination;
* Women with mental abnormal;
* Women did not cooperate or participate in other clinical trials;
* Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 2 years
  diagnostic accuracy comparison between Transvaginal Ultrasound diagnosis with and without Artificial Intelligence algorithm for ovarian cancer

SECONDARY OUTCOMES:
time cost for Transvaginal Ultrasound image interpretation | 2 years
  time cost for radiologists to interpret Transvaginal Ultrasound images

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD, PhD, Study Chair — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Yes
contact Prof. Gao for detailed study protocol or data after the study completed by e-mail
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after the study completed
Access Criteria: all investigators in this study field can contact Prof. Gao for access by e-mail